CLINICAL TRIAL: NCT01968031
Title: A Phase 3, 12-week, Double-Blind, Placebo-Controlled, Randomized, Multicenter Study to Evaluate the Efficacy of Oral Istradefylline 20 and 40 mg/Day as Treatment for Subjects With Moderate to Severe Parkinson's Disease
Brief Title: A 12-week Randomized Study to Evaluate Oral Istradefylline in Subjects With Moderate to Severe Parkinson's Disease
Acronym: KW-6002
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Collaborators: Kyowa Hakko Kirin Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6002-014; 2013-002254-70 (EudraCT Number)
Record Dates: First submitted 2013-10-18; First posted 2013-10-23 (Estimated); Results first posted 2020-11-20 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Idiopathic Parkinson's Disease
Keywords: Parkinson's disease; Moderate to Severe Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — istradefylline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Istradefylline 20 mg/day (Experimental): Istradefylline 20 mg and placebo to match istradefylline 40 mg:
  A daily, oral, double-blind treatment dose of both tablets will be taken in the morning for 12 weeks.
  Interventions: Drug: Istradefylline 20 mg; Drug: Placebo
- Istradefylline 40 mg/day (Experimental): Istradefylline 40 mg and placebo to match istradefylline 20 mg:
  A daily, oral, double-blind treatment dose of both tablets will be taken in the morning for 12 weeks.
  Interventions: Drug: Istradefylline 40 mg; Drug: Placebo
- Placebo (Placebo Comparator): Placebo to match istradefylline 20 mg and placebo to match istradefylline 40 mg:
  A daily, oral, double-blind treatment dose of both tablets will be taken in the morning for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Istradefylline 40 mg — Istradefylline 40 mg and placebo
  Other Names: KW-6002
  Arms: Istradefylline 40 mg/day
Drug: Istradefylline 20 mg — Istradefylline 20 mg and placebo
  Other Names: KW-6002
  Arms: Istradefylline 20 mg/day
Drug: Placebo — Placebo

SUMMARY:
This is a study to assess the efficacy and safety of oral Istradefylline (KW-6002) in patients with moderate to severe Parkinson's Disease. While on this study, participants will continue to take their usual, prescribed, stable regimen of Levodopa/Carbidopa or Levodopa/Benserazide therapy plus adjunct Parkinson's medications. Patients will be randomized 1:1:1 to receive either Istradefylline 20 mg per day, or Istradefylline 40 mg per day or an equivalent placebo. Patients will be treated for a 12 week period to demonstrate the effectiveness of Istradefylline in improving Parkinson's disease symptoms (referred to as improvement in patient OFF time) and that Istradefylline has an acceptable safety profile in this group.

ELIGIBILITY:
Inclusion Criteria:

* 30 years of age or older.
* UK Parkinson's Disease Society (UKPDS) brain bank criteria (Step 1 and 2) for PD
* PD Stages 2-4 in the ON state for Modified Hoehn and Yahr Scale.
* On levodopa therapy for at least 1 year with beneficial clinical response at the baseline visit
* Taking at least 400mg levodopa combination daily and on stable regimen of any other anti-Parkinsonian drugs (MAO-B, COMT, DA) for at least 2 weeks prior to randomization
* Stable dopaminergic regimen for at least 4 weeks immediately prior to randomization
* Documented end-of-dose wearing-off and levodopa-induced dyskinesia
* Have an average of two hours of OFF time per day

Exclusion Criteria:

* Subjects on apomorphine and/or dopamine receptor antagonists or direct gastrointestinal levodopa infusion.
* Subject who have had neurosurgical operation for PD
* Subjects taking A2a antagonist, potent CYP3A4 inhibitors, potent CYP34A inducers
* Subjects who smoke > 5 cigarettes/day

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 613 (Actual)
Dates: Start 2013-10; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyowa Hakko Kirin Pharma, Inc., Study Chair — Kyowa Hakko Kirin Pharma, Inc.
Locations (82):
- United States (39):
  - Kyowa PD Site, Phoenix, Arizona
  - Kyowa PD Site, Sun City, Arizona
  - Kyowa PD Site, Tucson, Arizona
  - Kyowa PD Site, Fountain Valley, California
  - Kyowa PD Site, Irvine, California
  - Kyowa PD Site, Los Angeles, California
  - Kyowa PD Site, Oxnard, California
  - Kyowa PD Site, Pasadena, California
  - Kyowa PD Site, Reseda, California
  - Kyowa PD Site, Sunnyvale, California
  - Kyowa PD Site, Torrance, California
  - Kyowa PD Site, Englewood, Colorado
  - Kyowa PD Site, Danbury, Connecticut
  - Kyowa PD Site, Boca Raton, Florida
  - Kyowa PD Site, Jacksonville, Florida
  - Kyowa PD Site, Panama City, Florida
  - Kyowa PD Site, Port Charlotte, Florida
  - Kyowa PD Site, Tampa, Florida
  - Kyowa PD Site, Atlanta, Georgia
  - Kyowa PD Site, Augusta, Georgia
  - Kyowa PD Site, Chicago, Illinois
  - Kyowa PD Site, Des Moines, Iowa
  - Kyowa PD Site, Kansas City, Kansas
  - Kyowa PD Site, Baltimore, Maryland
  - Kyowa PD Site, Boston, Massachusetts
  - Kyowa PD Site, West Bloomfield, Michigan
  - Kyowa PD Site, Minneapolis, Minnesota
  - Kyowa PD Site, St Louis, Missouri
  - Kyowa PD Site, Albany, New York
  - Kyowa PD Site, New York, New York
  - Kyowa PD Site, Asheville, North Carolina
  - Kyowa PD Site, Durham, North Carolina
  - Kyowa PD Site, Cincinnati, Ohio
  - Kyowa PD Site, Cleveland, Ohio
  - Kyowa PD Site, Toledo, Ohio
  - Kyowa PD Site, Philadelphia, Pennsylvania
  - Kyowa PD Site, Charleston, South Carolina
  - Kyowa PD Site, Dallas, Texas
  - Kyowa PD Site, Houston, Texas
- Canada (5):
  - Kyowa PD Site, Calgary, Alberta
  - Kyowa PD Site, Kingston, Ontario
  - Kyowa PD Site, Toronto, Ontario
  - Kyowa PD Site, Gatineau, Quebec
  - Kyowa PD Site, Québec, Quebec
- Czechia (4):
  - Kyowa PD Site, Brno
  - Kyowa PD Site, Litomyšl
  - Kyowa PD Site, Olomouc
  - Kyowa PD Site, Prague
- Germany (11):
  - Kyowa PD Site, Beelitz-Heilstätten
  - Kyowa PD Site, Berlin
  - Kyowa PD Site, Bremerhaven
  - Kyowa PD Site, Dresden
  - Kyowa PD Site, Göttingen
  - Kyowa PD Site, Haag
  - Kyowa PD Site, Kassel
  - Kyowa PD Site, Marburg
  - Kyowa PD Site, Munich
  - Kyowa PD Site, Tübingen
  - Kyowa PD Site, Ulm
- Israel (5):
  - Kyowa PD Site, Haifa
  - Kyowa PD Site, Jerusalem
  - Kyowa PD Site, Petach Tiqva
  - Kyowa PD Site, Ramat Gan
  - Kyowa PD Site, Tel Aviv
- Italy (8):
  - Kyowa PD Site, Cassino
  - Kyowa PD Site, Chieti
  - Kyowa PD Site, Grosseto
  - Kyowa PD Site, Pavia
  - Kyowa PD Site, Pisa
  - Kyowa PD Site, Rome
  - Kyowa PD Site, Venezia
  - Kyowa PD Site, Vicenza
- Poland (6):
  - Kyowa PD Site, Bydgoszcz
  - Kyowa PD Site, Kielce
  - Kyowa PD Site, Krakow
  - Kyowa PD Site, Lublin
  - Kyowa PD Site, Poznan
  - Kyowa PD Site, Warsaw
- Serbia (4):
  - Kyowa PD Site 1, Belgrade
  - Kyowa PD Site 2, Belgrade
  - Kyowa PD Site 4, Belgrade
  - Kyowa PD Site, Novi Sad

REFERENCES:
- See also: Fox Trial Finder is a clinical trial matching tool that helps a Parkinson's patient connect with research sites. Volunteers who sign up will receive a list of trials in their area. — https://foxtrialfinder.michaeljfox.org/trial/3633/

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo to match istradefylline 20 mg and placebo to match istradefylline 40 mg:
  A daily, oral, double-blind treatment dose of both tablets will be taken in the morning for 12 weeks.
  Placebo: Placebo
- Istradefylline 20 mg/Day: Istradefylline 20 mg and placebo to match istradefylline 40 mg:
  A daily, oral, double-blind treatment dose of both tablets will be taken in the morning for 12 weeks.
  Istradefylline 20 mg: Istradefylline 20 mg and placebo
  Placebo: Placebo
- Istradefylline 40 mg/Day: Istradefylline 40 mg and placebo to match istradefylline 20 mg:
  A daily, oral, double-blind treatment dose of both tablets will be taken in the morning for 12 weeks.
  Istradefylline 40 mg: Istradefylline 40 mg and placebo
  Placebo: Placebo
Period: Overall Study
Arm/Group | Placebo | Istradefylline 20 mg/Day | Istradefylline 40 mg/Day
Started | 204 | 202 | 207
Completed Week 2 | 197 | 190 | 199
Completed Week 6 | 191 | 183 | 187
Completed Week 10 | 187 | 181 | 181
Completed | 186 | 182 | 178
Not Completed | 18 | 20 | 29
Not completed — Adverse Event | 13 | 10 | 22
Not completed — Withdrawal by Subject | 3 | 7 | 3
Not completed — Did not meet entry criteria | 1 | 1 | 1
Not completed — Noncompliance | 0 | 0 | 2
Not completed — Failed inclusion criteria | 0 | 2 | 0
Not completed — Death | 0 | 0 | 1
Not completed — Prohibited concomitant medication | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Istradefylline 20 mg/Day | Istradefylline 40 mg/Day | Total
Number analyzed (Participants) | 204 | 201 | 207 | 612
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 104 | 108 | 101 | 313
  >=65 years | 100 | 93 | 106 | 299
Age, Continuous [Mean (Full Range); unit: years] | 63.8 [41 to 86] | 63.5 [41 to 87] | 64.5 [40 to 85] | 63.9 [40 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 76 | 81 | 237
  Male | 124 | 125 | 126 | 375
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 199 | 192 | 200 | 591
  Asian | 1 | 3 | 5 | 9
  Black or African American | 2 | 2 | 0 | 4
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Other - Filipino | 0 | 1 | 0 | 1
  Other - Hispanic | 0 | 1 | 0 | 1
  Other - Hispanic or Latino | 1 | 0 | 0 | 1
  Other - Indian | 1 | 0 | 0 | 1
  Other - Indian/Asian | 0 | 0 | 1 | 1
  Other - Puerto Rican | 0 | 0 | 1 | 1
  Other - did not wish to specify | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 11 | 11 | 10 | 32
  United States | 93 | 92 | 92 | 277
  Czechia | 22 | 23 | 23 | 68
  Poland | 24 | 23 | 23 | 70
  Italy | 21 | 18 | 20 | 59
  Israel | 11 | 12 | 12 | 35
  Serbia | 9 | 7 | 9 | 25
  Germany | 13 | 15 | 17 | 45

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Total Hours of Awake Time/Day Spent in the OFF State at Week 12
Description: Based on the 24-hour ON/OFF patient diary data.
Time Frame: Baseline, Week 2, Week 6, Week 10 and Week 12.
Population: The number of subjects in each row is based on the number of subjects with valid diary entries for the corresponding week
Measure: Median (Full Range); unit: hours
Arm/Group | Placebo | Istradefylline 20 mg/Day | Istradefylline 40 mg/Day
Number analyzed (Participants) | 198 | 194 | 200
hours
  Baseline | 5.17 [2.0 to 14.3] | 5.33 [1.0 to 12.2] | 4.92 [1.2 to 11.0]
  Week 2: number analyzed (Participants) | 198 | 193 | 200
  Week 2 | 4.83 [0.0 to 13.8] | 4.33 [0.0 to 11.5] | 4.08 [0.2 to 9.8]
  Week 6: number analyzed (Participants) | 192 | 184 | 190
  Week 6 | 4.17 [0.0 to 10.8] | 3.83 [0.0 to 9.5] | 3.83 [0.0 to 9.8]
  Week 10: number analyzed (Participants) | 187 | 179 | 176
  Week 10 | 4.33 [0.0 to 17.0] | 3.83 [0.0 to 11.3] | 3.50 [0.0 to 10.7]
  Week 12: number analyzed (Participants) | 188 | 179 | 200
  Week 12 | 4.17 [0.0 to 16.7] | 4.00 [0.0 to 11.3] | 3.83 [0.0 to 13.8]

2. Secondary Outcome: Total Hours of ON Time Per Day Without Troublesome Dyskinesia
Description: Based on Patient's ON/OFF Diary
Time Frame: Baseline, Week 2, Week 6, Week 10 and Week 12.
Population: as for outcome 1
Measure: Mean (Full Range); unit: hours
Arm/Group | Placebo | Istradefylline 20 mg/Day | Istradefylline 40 mg/Day
Number analyzed (Participants) | 198 | 194 | 200
hours
  Baseline | 9.22 [1.0 to 14.8] | 9.68 [1.8 to 15.0] | 9.72 [1.2 to 16.0]
  Week 2: number analyzed (Participants) | 198 | 193 | 200
  Week 2 | 9.89 [0.5 to 15.3] | 10.20 [0.0 to 16.8] | 10.46 [0.0 to 16.7]
  Week 6: number analyzed (Participants) | 192 | 184 | 190
  Week 6 | 10.18 [0.0 to 16.0] | 10.74 [0.0 to 17.0] | 10.46 [0.0 to 17.2]
  Week 10: number analyzed (Participants) | 187 | 179 | 181
  Week 10 | 10.12 [0.0 to 16.8] | 10.68 [0.0 to 16.2] | 10.53 [0.7 to 17.5]
  Week 12: number analyzed (Participants) | 188 | 179 | 176
  Week 12 | 10.13 [0.0 to 17.0] | 10.71 [0.0 to 17.8] | 10.53 [0.3 to 17.3]

3. Secondary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS) Motor Examination Score (Part III);
Description: The Unified Parkinson's Disease Rating Scale (UPDRS) evaluates various aspects of Parkinson's disease including non-motor and motor experiences of daily living and motor complications. Part III assesses the motor signs of Parkinson's Disease with a rating from 0 to 4, where 0 = normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe. The possible score range of Part III is 0 to 68. The lower the score, the more favorable the response.
Time Frame: Baseline, Week 2, Week 6, Week 10 and Week 12.
Population: The number of subjects in each row is based on the number of subjects with data for the corresponding week
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Placebo | Istradefylline 20 mg/Day | Istradefylline 40 mg/Day
Number analyzed (Participants) | 198 | 194 | 200
score on a scale
  Baseline | 22 [3 to 68] | 22.6 [4 to 62] | 23.5 [2 to 64]
  Week 2: number analyzed (Participants) | 197 | 192 | 200
  Week 2 | 20.1 [2 to 67] | 20.8 [2 to 61] | 20.7 [2 to 64]
  Week 6: number analyzed (Participants) | 197 | 188 | 196
  Week 6 | 19.9 [0 to 67] | 20.2 [0 to 61] | 20.2 [2 to 64]
  Week 10: number analyzed (Participants) | 189 | 184 | 181
  Week 10 | 19.2 [2 to 67] | 19.4 [0 to 60] | 19.9 [2 to 63]
  Week 12: number analyzed (Participants) | 188 | 181 | 178
  Week 12 | 19.4 [1 to 57] | 19.7 [0 to 60] | 19.6 [2 to 62]

4. Secondary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS) Activities of Daily Living (ADL) Score (Part II)
Description: The Unified Parkinson's Disease Rating Scale (UPDRS) evaluates various aspects of Parkinson's disease including non-motor and motor experiences of daily living and motor complications. Part II is a self-evaluation of the activities of daily life (ADL) including speech, swallowing, handwriting, dressing, hygiene, falling, salivating, turning in bed, walking, and cutting food with a rating from 0 to 4, where 0 = normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe. The possible score range of Part II is 0 to 52. The lower the score, the more favorable the response.
Time Frame: Baseline, Week 2, Week 6, Week 10 and Week 12.
Population: The number of subjects in each row is based on the number of subjects with data for the corresponding week
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Placebo | Istradefylline 20 mg/Day | Istradefylline 40 mg/Day
Number analyzed (Participants) | 198 | 194 | 200
score on a scale
  Baseline | 12.2 [0 to 27] | 12.0 [1 to 34] | 13.1 [0 to 32]
  Week 2 | 11.1 [1 to 27] | 10.7 [1 to 32] | 11.5 [0 to 32]
  Week 6: number analyzed (Participants) | 197 | 188 | 197
  Week 6 | 11.0 [0 to 27] | 10.5 [0 to 32] | 11.8 [0 to 32]
  Week 10: number analyzed (Participants) | 189 | 184 | 183
  Week 10 | 10.9 [0 to 27] | 10.8 [0 to 30] | 11.6 [0 to 31]
  Week 12: number analyzed (Participants) | 188 | 181 | 178
  Week 12 | 10.9 [0 to 27] | 10.7 [0 to 30] | 11.8 [0 to 30]

5. Secondary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS Mentation, Behaviour) and Mood (Part I)
Description: The Unified Parkinson's Disease Rating Scale (UPDRS) evaluates various aspects of Parkinson's disease including non-motor and motor experiences of daily living and motor complications. Part I is the evaluation of mentation, behavior, and mood with a rating from 0 to 4, where 0 = normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe. The possible score range of Part I is 0 to 16. The lower the score, the more favorable the response.
Time Frame: Baseline, Week 2, Week 6, Week 10 and Week 12.
Population: The number of subjects in each row is based on the number of subjects with data for the corresponding week
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Placebo | Istradefylline 20 mg/Day | Istradefylline 40 mg/Day
Number analyzed (Participants) | 198 | 194 | 200
score on a scale
  Baseline | 1.8 [0 to 7] | 1.3 [0 to 7] | 1.7 [0 to 9]
  Week 2 | 1.4 [0 to 9] | 1.1 [0 to 5] | 1.3 [0 to 8]
  Week 6: number analyzed (Participants) | 197 | 188 | 197
  Week 6 | 1.5 [0 to 7] | 1.3 [0 to 6] | 1.5 [0 to 7]
  Week 10: number analyzed (Participants) | 189 | 184 | 183
  Week 10 | 1.5 [0 to 7] | 1.4 [0 to 8] | 1.4 [0 to 6]
  Week 12: number analyzed (Participants) | 188 | 181 | 178
  Week 12 | 1.5 [0 to 7] | 1.4 [0 to 8] | 1.4 [0 to 6]

6. Secondary Outcome: Total UPDRS (Parts I + II + III);
Description: The Unified Parkinson's Disease Rating Scale (UPDRS) evaluates various aspects of Parkinson's disease including non-motor and motor experiences of daily living and motor complications with a rating from 0 to 4, where 0 = normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe. The total possible score range for all parts combined is 0 to 136. The lower the score, the more favorable the response.
Time Frame: Baseline, Week 2, Week 6, Week 10 and Week 12.
Population: The number of subjects in each row is based on the number of subjects with data for the corresponding week
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Placebo | Istradefylline 20 mg/Day | Istradefylline 40 mg/Day
Number analyzed (Participants) | 198 | 194 | 200
score on a scale
  Baseline | 35.9 [10 to 98] | 35.9 [9 to 102] | 38.3 [8 to 102]
  Week 2: number analyzed (Participants) | 197 | 192 | 200
  Week 2 | 32.6 [8 to 96] | 32.7 [5 to 98] | 33.6 [4 to 102]
  Week 6: number analyzed (Participants) | 197 | 188 | 196
  Week 6 | 32.4 [3 to 96] | 31.9 [3 to 98] | 33.5 [4 to 102]
  Week 10: number analyzed (Participants) | 189 | 184 | 181
  Week 10 | 31.6 [6 to 96] | 31.6 [2 to 93] | 33.0 [5 to 100]
  Week 12: number analyzed (Participants) | 188 | 181 | 178
  Week 12 | 31.9 [7 to 86] | 31.9 [1 to 93] | 32.9 [5 to 98]

7. Secondary Outcome: Patient Global Impression - Improvement (PGI-I) Scale
Description: The "key symptom" on the PGI-I was evaluated at baseline and subsequent post-baseline visits for the subject's overall condition and the symptoms of fatigue, sleep, motivation to get things done, and each subject's key symptom. Subjects rated each on a scale of 1 to 5 for change from baseline utilizing the following scale:
  * 1 = Moderate improvement (or greater)
  * 2 = Mild improvement
  * 3 = No change from baseline
  * 4 = Mild deterioration
  * 5 = Moderate deterioration (or greater)
  A lower number is a better outcome. Overall condition is presented below.
Time Frame: Baseline, Week 2, Week 6, Week 10, Week 12 and 30-day FU visit
Population: The number of subjects in each row is based on the number of subjects with data for the corresponding week
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Istradefylline 20 mg/Day | Istradefylline 40 mg/Day
Number analyzed (Participants) | 198 | 194 | 200
Participants
  Week 2: number analyzed (Participants) | 198 | 193 | 199
  Week 2: 1 = Moderate improvement (or greater) | 20 | 26 | 20
  Week 2: 2 = Mild improvement | 73 | 80 | 68
  Week 2: 3 = No change from baseline | 87 | 68 | 94
  Week 2: 4 = Mild deterioration | 15 | 13 | 15
  Week 2: 5 = Moderate deterioration (or greater) | 3 | 6 | 2
  Week 6: number analyzed (Participants) | 197 | 187 | 197
  Week 6: 1 = Moderate improvement (or greater) | 31 | 37 | 35
  Week 6: 2 = Mild improvement | 61 | 65 | 56
  Week 6: 3 = No change from baseline | 83 | 63 | 66
  Week 6: 4 = Mild deterioration | 21 | 19 | 37
  Week 6: 5 = Moderate deterioration (or greater) | 1 | 3 | 3
  Week 10: number analyzed (Participants) | 189 | 183 | 183
  Week 10: 1 = Moderate improvement (or greater) | 28 | 33 | 32
  Week 10: 2 = Mild improvement | 66 | 63 | 57
  Week 10: 3 = No change from baseline | 68 | 58 | 65
  Week 10: 4 = Mild deterioration | 22 | 22 | 24
  Week 10: 5 = Moderate deterioration (or greater) | 5 | 7 | 5
  Week 12: number analyzed (Participants) | 188 | 181 | 177
  Week 12: 1 = Moderate improvement (or greater) | 32 | 38 | 29
  Week 12: 2 = Mild improvement | 59 | 62 | 60
  Week 12: 3 = No change from baseline | 72 | 52 | 59
  Week 12: 4 = Mild deterioration | 20 | 26 | 23
  Week 12: 5 = Moderate deterioration (or greater) | 5 | 3 | 6
  30-Day Follow Up: number analyzed (Participants) | 46 | 51 | 56
  30-Day Follow Up: 1 = Moderate improvement (or greater) | 3 | 1 | 3
  30-Day Follow Up: 2 = Mild improvement | 10 | 3 | 7
  30-Day Follow Up: 3 = No change from baseline | 22 | 21 | 28
  30-Day Follow Up: 4 = Mild deterioration | 9 | 14 | 16
  30-Day Follow Up: 5 = Moderate deterioration (or greater) | 2 | 12 | 2

8. Secondary Outcome: Sleep Time in Hours Per Day Based Upon 24-hour Diaries.
Time Frame: Baseline, Week 2, Week 6, Week 10 and Week 12.
Population: as for outcome 1
Measure: Mean (Full Range); unit: hours
Arm/Group | Placebo | Istradefylline 20 mg/Day | Istradefylline 40 mg/Day
Number analyzed (Participants) | 198 | 194 | 200
hours
  Baseline | 8.11 [2.2 to 15.7] | 8.04 [3.7 to 13.2] | 8.11 [3.0 to 14.0]
  Week 2: number analyzed (Participants) | 198 | 193 | 200
  Week 2 | 8.10 [4.0 to 14.0] | 8.14 [2.8 to 15.3] | 8.13 [3.5 to 14.8]
  Week 6: number analyzed (Participants) | 192 | 184 | 190
  Week 6 | 8.23 [4.3 to 12.5] | 8.21 [3.0 to 15.5] | 8.40 [3.8 to 16.8]
  Week 10: number analyzed (Participants) | 187 | 179 | 181
  Week 10 | 8.38 [3.7 to 13.7] | 8.30 [2.8 to 14.5] | 8.44 [4.3 to 14.2]
  Week 12: number analyzed (Participants) | 188 | 179 | 176
  Week 12 | 8.26 [2.3 to 12.7] | 8.13 [3.2 to 14.2] | 8.30 [3.8 to 15.0]

9. Secondary Outcome: Percentage of Awake Time Per Day Spent in the OFF State
Time Frame: Baseline, Week 2, Week 6, Week 10 and Week 12.
Population: as for outcome 1
Measure: Mean (Full Range); unit: percentage of hours
Arm/Group | Placebo | Istradefylline 20 mg/Day | Istradefylline 40 mg/Day
Number analyzed (Participants) | 198 | 194 | 200
percentage of hours
  Baseline | 34.55 [12.7 to 84.4] | 33.92 [7.1 to 82.1] | 33.16 [8.2 to 72.2]
  Week 2: number analyzed (Participants) | 198 | 193 | 200
  Week 2 | 30.95 [0.0 to 93.2] | 29.46 [0.0 to 76.0] | 27.45 [1.0 to 60.2]
  Week 6: number analyzed (Participants) | 192 | 184 | 190
  Week 6 | 28.04 [0.0 to 76.5] | 26.31 [0.0 to 76.4] | 26.39 [0.0 to 63.9]
  Week 10: number analyzed (Participants) | 187 | 179 | 181
  Week 10 | 28.80 [0.0 to 89.2] | 25.69 [0.0 to 75.3] | 25.09 [0.0 to 65.6]
  Week 12: number analyzed (Participants) | 188 | 179 | 176
  Week 12 | 28.62 [0.0 to 92.9] | 26.24 [0.0 to 85.2] | 26.51 [0.0 to 74.5]

10. Secondary Outcome: Percentage of ON Time Per Day Without Troublesome Dyskinesia.
Time Frame: Baseline, Week 2, Week 6, Week 10 and Week 12.
Population: as for outcome 1
Measure: Mean (Full Range); unit: percentage of hours
Arm/Group | Placebo | Istradefylline 20 mg/Day | Istradefylline 40 mg/Day
Number analyzed (Participants) | 198 | 194 | 200
percentage of hours
  Baseline | 58.54 [5.4 to 85.2] | 61.04 [11.5 to 86.0] | 61.54 [6.9 to 91.8]
  Week 2: number analyzed (Participants) | 198 | 193 | 200
  Week 2 | 62.99 [2.7 to 100.0] | 64.72 [0.0 to 100.0] | 66.26 [0.0 to 96.7]
  Week 6: number analyzed (Participants) | 192 | 184 | 190
  Week 6 | 65.34 [0.0 to 99.0] | 68.51 [0.0 to 98.8] | 67.55 [0.0 to 100.0]
  Week 10: number analyzed (Participants) | 187 | 179 | 181
  Week 10 | 65.33 [0.0 to 100.0] | 68.65 [0.0 to 100.0] | 68.17 [4.4 to 100.0]
  Week 12: number analyzed (Participants) | 188 | 179 | 176
  Week 12 | 65.17 [0.0 to 100.0] | 68.17 [0.0 to 100.0] | 67.64 [2.0 to 100.0]

11. Secondary Outcome: Montreal Cognitive Assessment (MoCA)
Description: The Montreal Cognitive Assessment (MoCA) assesses different cognitive domains, broken down as follows:
  Visuospatial and executive functioning: 5 points Animal Naming: 3 points Attention: 6 points Language: 3 points Abstraction: 2 points Delayed recall (short-term memory): 5 points Orientation: 6 points
  Scores can range from 0 to 30. A score of 26 or above is considered normal.
Time Frame: Baseline and Week 12.
Population: Intent-to-Treat Analysis set: Includes all subjects randomized to a treatment arm and with both a valid baseline and at least one valid post-baseline patient diary.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Placebo | Istradefylline 20 mg/Day | Istradefylline 40 mg/Day
Number analyzed (Participants) | 198 | 194 | 200
score on a scale
  Score at Baseline | 28 [26 to 30] | 28 [26 to 30] | 28 [26 to 30]
  Score at Week 12 | 27.8 [19 to 30] | 27.9 [18 to 30] | 27.7 [20 to 30]

12. Secondary Outcome: Beck Depression Inventory (BDI)
Description: The Beck Depression Inventory is a 21-question test that measures the severity of depression. Subjects rated each on a scale of 0 to 3 for change from baseline utilizing the following scale:
  * 0 = I do not feel sad
  * 1 = I feel sad
  * 2 = I am sad all the time and I can't snap out of it
  * 3 = I am so sad or unhappy that I can't stand it
  The test is scored for each question using the above scale to determine the severity of depression. Scoring is as shown below:
  * 0 to 9: minimal depression
  * 10 to 18: mild depression
  * 19 to 29: moderate depression
  * 30 to 63: severe depression
Time Frame: Baseline and Week 12.
Population: The number of subjects in each row is based on the number of subjects with data for the corresponding week
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Placebo | Istradefylline 20 mg/Day | Istradefylline 40 mg/Day
Number analyzed (Participants) | 198 | 194 | 199
score on a scale
  Baseline: number analyzed (Participants) | 198 | 194 | 198
  Baseline | 8.8 [0 to 20] | 8.6 [0 to 28] | 9.3 [0 to 20]
  Week 12: number analyzed (Participants) | 198 | 191 | 199
  Week 12 | 7.9 [0 to 28] | 7.5 [0 to 27] | 8.3 [0 to 32]

ADVERSE EVENTS:
Arm/Group | Placebo | Istradefylline 20 mg/Day | Istradefylline 40 mg/Day
All-Cause Mortality (participants affected / at risk) | 0/204 | 0/201 | 1/207
Serious Adverse Events (participants affected / at risk) | 7/204 | 6/201 | 8/207
Other Adverse Events (participants affected / at risk) | 111/204 | 117/201 | 132/207
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=204) | Istradefylline 20 mg/Day (N=201) | Istradefylline 40 mg/Day (N=207)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Mitral valve prolapse (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis syndrome (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Anaesthetic complication neurological (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Medical observation (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Parkinson's disease (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=204) | Istradefylline 20 mg/Day (N=201) | Istradefylline 40 mg/Day (N=207)
Anaemia (Blood and lymphatic system disorders) | 3 (4) | 2 (2) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Heart alternation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Left ventricular hypertrophy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 2 (2)
Presbyacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Cerumen impaction (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Myopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 2 (2)
Binocular eye movement disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vitreous detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3) | 6 (6)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 8 (8) | 12 (13)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Faecal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 5 (5) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 8 (8) | 1 (1) | 4 (5)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (3)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (3) | 8 (8)
Intestinal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Anal spasm (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Irritability (General disorders) | 2 (2) | 1 (1) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 6 (6) | 3 (3) | 8 (8)
Energy increased (General disorders) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1) | 2 (2)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 1 (1)
Therapeutic response decreased (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 2 (2) | 1 (1)
Suprapubic pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 3 (3) | 3 (3) | 2 (2)
Oedema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 2 (2) | 0 (0) | 4 (4)
Vessel puncture site bruise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Local swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (2)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 6 (7) | 6 (6) | 7 (8)
Tooth abscess (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Tinea pedis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 3 (3)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (2) | 8 (10) | 2 (2)
Nail infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lyme disease (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 4 (4) | 4 (4)
Croup infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 6 (6) | 2 (2) | 3 (3)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 3 (3) | 2 (2)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Suture rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 3 (3)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Periorbital contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lip injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (4)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 9 (12) | 13 (17) | 18 (22)
Sternal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 4 (4) | 4 (5)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Corneal abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 5 (5) | 3 (5)
Blood calcium increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood calcium decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 0 (0) | 1 (2)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Biopsy skin (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (2) | 2 (2) | 1 (1)
Amylase increased (Investigations) | 4 (4) | 2 (2) | 2 (3)
White blood cells urine positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 1 (2) | 1 (1) | 1 (1)
Weight increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 3 (3) | 2 (2)
Urine transitional cells present (Investigations) | 1 (1) | 0 (0) | 0 (0)
Urine ketone body present (Investigations) | 1 (1) | 0 (0) | 0 (0)
Urinary casts (Investigations) | 0 (0) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Specific gravity urine increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Red blood cell count decreased (Investigations) | 0 (0) | 2 (2) | 0 (0)
QRS axis abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Protein urine present (Investigations) | 1 (1) | 0 (0) | 0 (0)
Precancerous cells present (Investigations) | 1 (1) | 0 (0) | 0 (0)
Occult blood (Investigations) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Monocyte count increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Nitrite urine present (Investigations) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte percentage decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (2) | 0 (0) | 1 (2)
Lipase increased (Investigations) | 5 (5) | 2 (2) | 2 (3)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Heart rate increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 1 (1) | 1 (1)
Haematocrit decreased (Investigations) | 1 (1) | 2 (2) | 0 (0)
Red blood cells urine positive (Investigations) | 1 (1) | 0 (0) | 1 (1)
Eosinophil percentage increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Eosinophil count increased (Investigations) | 1 (1) | 0 (0) | 2 (2)
Electrocardiogram abnormal (Investigations) | 2 (2) | 0 (0) | 1 (1)
Crystal urine present (Investigations) | 1 (1) | 1 (1) | 1 (2)
Cardiac murmur (Investigations) | 1 (1) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 1 (1) | 2 (2) | 1 (1)
Blood triglycerides increased (Investigations) | 3 (3) | 2 (2) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Blood uric acid increased (Investigations) | 0 (0) | 3 (3) | 2 (2)
Blood potassium increased (Investigations) | 2 (2) | 0 (0) | 1 (1)
Blood phosphorus decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 3 (3) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 3 (3)
Blood urine present (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 5 (5) | 3 (3) | 3 (3)
Blood cholesterol increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Lactose intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperphagia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (3)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0) | 3 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 2 (2)
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myosclerosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Posture abnormal (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Facial asymmetry (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Bone disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 2 (2)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (7) | 4 (4) | 5 (5)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Speech disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 5 (5) | 4 (4) | 5 (5)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Psychomotor hyperactivity (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Postural reflex impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Poor quality sleep (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Parkinson's disease (Nervous system disorders) | 2 (2) | 2 (2) | 2 (2)
Paraesthesia (Nervous system disorders) | 1 (1) | 7 (7) | 5 (5)
Nerve root compression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Nerve compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Micrographia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Meralgia paraesthetica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Mental impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
On and off phenomenon (Nervous system disorders) | 9 (10) | 2 (2) | 6 (6)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Intercostal neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 5 (5) | 4 (4) | 4 (4)
Freezing phenomenon (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2)
Dystonia (Nervous system disorders) | 0 (0) | 1 (1) | 2 (3)
Dyskinesia (Nervous system disorders) | 14 (14) | 23 (30) | 34 (37)
Sciatica (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 2 (2) | 3 (3) | 2 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 5 (5) | 6 (6) | 9 (11)
Disturbance in attention (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Bradykinesia (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1)
Akinesia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Apathy (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 3 (3) | 2 (2) | 5 (6)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 1 (1) | 4 (4)
Terminal insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 3 (3) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1) | 2 (2) | 1 (1)
Rapid eye movements sleep abnormal (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2)
Paranoia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Mood altered (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Middle insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Mania (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Libido increased (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 5 (6) | 10 (10) | 7 (7)
Initial insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Impulse-control disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Illusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Hypomania (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Hypersexuality (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Hallucination, visual (Psychiatric disorders) | 2 (2) | 2 (2) | 0 (0)
Hallucination, auditory (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Hallucination (Psychiatric disorders) | 2 (2) | 1 (1) | 4 (5)
Depression (Psychiatric disorders) | 2 (2) | 3 (3) | 2 (2)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Delusion (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urge incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Nephritis (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 2 (2) | 0 (0) | 2 (2)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Azotaemia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Breast tenderness (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rales (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (4) | 3 (3)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 3 (3)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Livedo reticularis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Raynaud's phenomenon (Vascular disorders) | 0 (0) | 1 (2) | 0 (0)
Peripheral coldness (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (2) | 7 (8) | 3 (3)
Orthostatic hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 3 (3) | 2 (2) | 0 (0)
Hypoperfusion (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 4 (5)
Hot flush (Vascular disorders) | 1 (1) | 3 (3) | 2 (2)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Blood pressure fluctuation (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Accelerated hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days